CLINICAL TRIAL: NCT01918852
Title: S1 Versus Capecitabine in the First Line Treatment of Metastatic Colorectal Cancer Patients, the SALTO Randomised Phase III Study of the Dutch Colorectal Cancer Group. A Safety Evaluation of Oral Fluoropyrimidines
Brief Title: S-1 Versus Capecitabine in the First Line Treatment of MCC Patients.
Acronym: SALTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALTO
Record Dates: First submitted 2013-06-24; First posted 2013-08-08 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Metastases
Keywords: Hand-foot syndrome; Toxicity; Fluoropyrimidine; Capecitabine; Teysuno; S1
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Hand-Foot Syndrome | interventions — Capecitabine; tegafur-gimeracil-oteracil; S 1 (combination); Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine (Active Comparator): Capecitabine 1250 mg/m2 for patients < 70 years of age, and 1000 mg/m2 for patients ≥ 70 years of age, orally b.i.d. day 1-14 with or without bevacizumab 7.5 mg/kg i.v. day 1.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab
- S1 (Experimental): S-1 30 mg/m2 orally b.i.d. irrespective of age, day 1-14 with or without bevacizumab 7.5 mg/kg i.v. day 1.
  Interventions: Drug: Teysuno; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
  Arms: Capecitabine
Drug: Teysuno
  Other Names: S1
  Arms: S1
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The study is a two-arm randomised phase III trial. Patients will be randomised to receive capecitabine (arm A) or S-1 (arm B). Bevacizumab may be added according to the choice of the investigator. Patients will be followed 3-weekly at the outpatient clinic, toxicity will be assessed according to study protocol guidelines. Patients will be evaluated every 3 cycles for response. Upon disease progression patients will be treated according to the local investigators

DETAILED DESCRIPTION:
Capecitabine, an oral fluoropyrimidine, has shown a comparable efficacy but a better tolerability compared to bolus 5-FU/LV. However, capecitabine has a higher incidence of hand-foot syndrome (HFS). HFS is characterized by erythema, dysesthesia and/or paresthesia of the palms of the hands or soles of feet. In advanced stage, desquamation, ulceration and blistering can occur. Although HFS is not life threatening, it can cause significant discomfort and impairment of function, especially in elderly patients. This adverse event is becoming particularly relevant since many patients may require the administration of capecitabine over prolonged periods of time.

S-1 (Teysuno®) is an oral fluoropyrimidine that has shown comparable efficacy to 5FU and capecitabine in gastrointestinal cancers but is associated with a much lower incidence of HFS. Studies on S-1 have mainly been performed in Asian patients,which population has known differences in tumour biology and toxicity compared to Western population. S-1 has shown comparable efficacy to other fluoropyrimidines as monotherapy or in combination chemotherapy schedules in several gastrointestinal tumors. However, given the lack of data from prospective studies on S-1 as monochemotherapy in metastatic colorectal cancer in Western patients, this study is designed to compare S-1 and capecitabine monotherapy in terms of safety, with particular interest in HFS, in metastatic colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer.
* Distant metastases (patients with only local recurrence are not eligible).
* Unidimensionally measurable disease (≥1 cm on spiral CT scan or ≥2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation.
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.
* Age ≥ 18 years
* Planned treatment with fluoropyrimidine monotherapy with or without bevacizumab.
* WHO performance status 0-2 (Karnofsky PS ≥70%)
* Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥1.5 x 109/L, platelets ≥ 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, ≥30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases).
* Life expectancy > 12 weeks.
* Negative pregnancy test in women with childbearing potential.
* Expected adequacy of follow-up.
* Institutional Review Board approval.
* Written informed consent.

Exclusion Criteria:

* Prior adjuvant treatment for stage II/III colorectal cancer completed within 6 months prior to randomisation.
* Any prior adjuvant treatment after resection of distant metastases.
* Any previous systemic treatment for metastatic disease.
* History or clinical signs/symptoms of CNS metastases.
* History of a second malignancy <5 years with the exception of adequately treated carcinoma of cervix or basal/squamous cell carcinoma of skin.
* Previous intolerance of capecitabine.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency or treatment within 4 weeks with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine.
* Planned radical resection of metastases after downsizing by systemic treatment.
* Significant cardiovascular disease < 1 yr before randomisation (symptomatic congestive heart failure, myocardial ischemia or infarction, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, arterial thrombosis, cerebrovascular event, pulmonary embolism).
* Any significant cardiovascular events during previous fluoropyrimidine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence of HFS in first line treatment | HFS will be assessed every 3 weeks up to 6 months average.
  To determine the incidence of HFS in first line treatment with S-1 compared to capecitabine in patients with metastatic colorectal cancer.

SECONDARY OUTCOMES:
Grade 3 HFS | HFS will be assessed every 3 weeks, up to 6 months average
  Incidence of grade 3 hand-foot syndrome, according to CTC 4.0.
Progression-free survival | Every 9 weeks, for 6 months (average)
  Time from randomisation until progression or death whichever comes first
Overall toxicity | Every 3 weeks, for 6 months (average)
  Adverse events graded accoording to the NCI CTCAE version 4
Overall survival | 2 years
  From date of randomisation to death or last known to be alive
Response rate | Response will be assessed every 9 weeks, up to 6 months average.
  Response acccording to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis JA Punt, Prof MD PhD, Principal Investigator — Amsterdam Medical Centre
Locations (24):
- Netherlands (24):
  - Medisch Centrum Alkmaar, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Nederlands Kanker Instituut/Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Academic Medical Centre, Amsterdam
  - OLVG, Amsterdam
  - VUMC, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Ziekenhuis Lievensberg, Bergen op Zoom
  - Amphia Ziekenhuis, Breda
  - Slingeland Ziekenhuis, Doetinchem
  - Catherina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - St Jansdal, Harderwijk
  - Spaarne Ziekenhuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Antonius Ziekenhuis, Nieuwegein
  - Waterland Ziekenhuis, Purmerend
  - Sint Franciscus Gasthuis, Rotterdam
  - Vlietland Ziekenhuis, Schiedam
  - Orbis Medisch Centrum, Sittard
  - Tweesteden Ziekenhuis, Tilburg
  - University Medical Centre Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Zaans Medisch Centrum, Zaandam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwakman JJM, van Werkhoven E, Simkens LHJ, van Rooijen JM, van de Wouw YAJ, Tije AJT, Creemers GM, Hendriks MP, Los M, van Alphen RJ, Polee MB, Muller EW, van der Velden AMT, van Voorthuizen T, Koopman M, Mol L, Punt CJA. Updated Survival Analysis of the Randomized Phase III Trial of S-1 Versus Capecitabine in the First-Line Treatment of Metastatic Colorectal Cancer by the Dutch Colorectal Cancer Group. Clin Colorectal Cancer. 2019 Jun;18(2):e229-e230. doi: 10.1016/j.clcc.2019.01.002. Epub 2019 Jan 29. No abstract available. PMID 30782413
- [Derived] Kwakman JJM, Simkens LHJ, van Rooijen JM, van de Wouw AJ, Ten Tije AJ, Creemers GJM, Hendriks MP, Los M, van Alphen RJ, Polee MB, Muller EW, van der Velden AMT, van Voorthuizen T, Koopman M, Mol L, van Werkhoven E, Punt CJA. Randomized phase III trial of S-1 versus capecitabine in the first-line treatment of metastatic colorectal cancer: SALTO study by the Dutch Colorectal Cancer Group. Ann Oncol. 2017 Jun 1;28(6):1288-1293. doi: 10.1093/annonc/mdx122. PMID 28383633
- See also: Related Info — http://www.dccg.nl